CLINICAL TRIAL: NCT06631352
Title: Outcomes and Prognostic Factors in Hepatopancreatoduodenectomy
Acronym: HPD_single
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Young Jang, Professor, Seoul National University Hospital
Other Study IDs: 2407-049-1551
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-05

CONDITIONS: Hepatopancreaticobiliary (HPB) Malignancy; Gall Bladder Cancer; Bile Duct Cancer; Pancreatoduodenectomy; Hepatectomy
Keywords: Hepatopancreatoduodenectomy
MeSH Terms: conditions — Neoplasms; Gallbladder Neoplasms; Bile Duct Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GB cancer: Patients who were diagnosed with gallbladder cancer and underwent the hepatopancreatoduodenectomy.
  Interventions: Other: Hepatopancreatoduodenectomy
- CCA: Patients who were diagnosed with cholangiocarcinoma and underwent the hepatopancreatoduodenectomy.
  Interventions: Other: Hepatopancreatoduodenectomy

INTERVENTIONS:
Other: Hepatopancreatoduodenectomy — Pancreatoduodenectomy with liver resection

SUMMARY:
1. In biliary tract malignancies, achieving a microscopically clear resection margin (R0) is considered the only treatment for a cure.
2. Hepatopancreatoduodenectomy(HPD) has been considered a surgical option for patients with extensive bile duct or gallbladder cancer to achieve an R0 resection.
3. The associated high morbidity and mortality rates have prevented HPD from becoming a standard surgical procedure worldwide.
4. Over the past few decades, the understanding of the bile duct anatomy has significantly improved, and many methods have been developed to assess liver function and future remnant liver volume.
5. We aimed to evaluate the short- and long-term outcomes of HPD and to assess risk factors associated with survival, early recurrence, and major complications to better evaluate the potential of the procedure as a standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received hepatopancreatoduodenectomy between January 2000 and December 2023.

Exclusion Criteria:

* Patients who had R2 resection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included 51 patients who underwent HPD at Seoul National University Hospital between January 2000 and December 2023. One patient who had an R2 resection was excluded from the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
5-year overall survival | assessed up to 60months
  the time from the date of surgery to the date of death or last follow-up.
5-year disease-free survival | assessed up to 60months
  from the date of surgery to the first instance of recurrence, death, or last follow-up date.

SECONDARY OUTCOMES:
Post operative complications | assessed up to 30 days from the surgery
  Complications occured after the HPD. For example, there are post-hepatectomy liver failure, postoperative pancreatic fistula, ileus, fluid collection, pleural effusion, and etc.